CLINICAL TRIAL: NCT05624099
Title: Prospective Single-arm, Exploratory, Multicenter Phase II Clinical Study of Camrelizumab Combined With Chemoradiotherapy in the Treatment of Advanced First-line Esophageal Phosphorous Carcinoma
Brief Title: Camrelizumab Combined With Chemoradiotherapy in Advanced Esophageal Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Advanced immunotherapy CRT
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Neoplasms; Esophageal Diseases; Digestive System Neoplasms
Keywords: Immunotherapy; Platinum; radiotherapy; Paclitaxel
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases; Digestive System Neoplasms | interventions — camrelizumab; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- drug (Experimental): 1. camrelizumab 200mg intravenous drip d1q3w
  2. Paclitaxel: 150mg/m2 d1 q3w
  3. Platinum: Cisplatin, carboplatin, nedaplatin and other platinum drugs
  4. Radiotherapy dose: 5040cGy/28f radiotherapy efficacy evaluation after 2-3 cycles of chemotherapy PR/SD received local radiotherapy.
  Interventions: Drug: camrelizumab; Drug: Paclitaxel drugs; Drug: Platinum drug; Radiation: Radiation

INTERVENTIONS:
Drug: camrelizumab — 200mg intravenous drip d1q3w
Drug: Paclitaxel drugs — 150mg/m2 d1 q3w
Drug: Platinum drug — Cisplatin, carboplatin, nedaplatin and other platinum drugs
Radiation: Radiation — Dose: 5040cGy/28f

SUMMARY:
This is a prospective single-arm exploratory clinical study. The efficacy and safety of camrelizumab combined with chemoradiotherapy and camrelizumab combined with chemotherapy were evaluated in patients with advanced esophageal cancer who had not previously received any systemic antitumor therapy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent and voluntarily participate in this study;
2. Patients with esophageal squamous cell carcinoma confirmed by histopathology and/or immunohistochemistry (8th edition 2017) had UICC/AJCC TNM stage IVA or oligometastatic stage IVB;
3. Survival is expected to exceed 3 months
4. Age 18-75;
5. ECOG PS 0-2
6. Never received any systemic anti-tumor therapy for esophageal cancer, including radiotherapy, chemotherapy, targeted and immunotherapy;
7. Have at least one measurable lesion
8. Normal function of major organs, including:

   1. Routine blood test (no blood components, cell growth factors, whitening drugs, platelet raising drugs, and anemia correcting drugs are allowed within 14 days before the first use of study drugs)

      White blood cell count ≥ 3.0×10^9/L

      Neutrophil count ≥ 1.0×10^9/L

      Platelet count ≥ 80×109/L

      Hemoglobin ≥ 80 g/L
   2. Blood biochemical examination:

   Total bilirubin ≤ 1.5×ULN

   ALT ≤2.5×ULN, AST ≤2.5×ULN,

   Serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 45mL/min
9. Subjects have good compliance and cooperate with follow-up

Exclusion Criteria:

1. The presence of uncontrollable pleural effusion, pericardial effusion or ascites that require repeated drainage;
2. Poor nutritional status, BMI < 18.5 Kg/m^2; If symptomatic nutritional support was corrected before randomization, enrollment could be considered after evaluation by the principal investigator;
3. Gastrointestinal bleeding (bleeding volume > 200ml/ day);
4. Patients with deep ulcers as determined by the investigator;
5. Previous allergy to monoclonal antibodies, any component of camrelizumab, paclitaxel, cisplatin or other platinum-based drugs;
6. Has received or is receiving any of the following medical treatment:

   1. any radiation, chemotherapy or other antitumor drugs for the tumor;
   2. Being treated with immunosuppressive agents or systemic hormones for immunosuppression purposes (dose >10mg/ day prednisone or equivalent) within 2 weeks prior to the first use of the study drug; In the absence of active autoimmune disease, inhaled or topical steroids and adrenocorticosteroid replacement at a dose of >10mg/ day or its equivalent are permitted;
   3. Received live attenuated vaccine within 4 weeks before the first administration of the study drug;
   4. Major surgery or severe trauma within 4 weeks before the first use of the study drug;
7. A history of any active autoimmune disease or autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (which may be considered for inclusion after hormone replacement therapy); Patients with complete remission of psoriasis or childhood asthma/allergies who did not require any intervention as adults were considered for inclusion, but patients requiring medical intervention with bronchodilators were not included;
8. A history of immunodeficiency, including being HIV positive, or suffering from another acquired or congenital immunodeficiency disease, or a history of organ transplantation or allogeneic bone marrow transplantation;
9. The presence of poorly controlled cardiac clinical symptoms or diseases, including but not limited to:

   Such as (1) NYHAII grade or above heart failure; (2) unstable angina pectoris; (3) myocardial infarction occurred within 1 year; (4) Clinically significant supraventricular or ventricular arrhythmias are not well controlled without clinical intervention or after clinical intervention;
10. Severe infection (CTCAE > 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia, infection complications requiring hospitalization; Baseline chest imaging examination indicated active pulmonary inflammation, signs and symptoms of infection within 14 days before the first use of study drugs, or the need for oral or intravenous antibiotic treatment, except for prophylactic antibiotic use;
11. Patients with active pulmonary tuberculosis infection found by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or with a history of active pulmonary tuberculosis infection more than 1 year ago but without regular treatment;
12. The presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL) and hepatitis C (HCV antibody positive and HCV RNA above the assay limit);
13. In the judgment of the investigator, there are other factors that may lead to the forced termination of the study, such as the presence of other serious medical conditions (including mental illness) requiring concomitant treatment, alcoholism, substance abuse, family or social factors, and factors that may affect the safety or compliance of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | 3 years
  ORR is determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  Defined as the time from the enrollment to death from any cause
Progression free survival(PFS) | 3 years
  It is defined as the time from enrollment to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, China

IPD SHARING:
Plan to Share IPD: Undecided